CLINICAL TRIAL: NCT01756716
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Effect on Urine Albumin-to-Creatinine Ratio (UACR), Pharmacodynamics, Safety, Tolerability and Pharmacokinetics of Multiple Oral Doses of MT-3995 as Add-on Therapy to ACE-I or ARB in Type II Diabetic Nephropathy Subjects With Albuminuria and an eGFR ≥30-<60 mL/Min/1.73m^2
Brief Title: A Study to Evaluate Pharmacodynamics, Safety, Tolerability and Pharmacokinetics of MT-3995 in Type II Diabetic Nephropathy Subjects With Albuminuria and Moderately Decreased GFR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-3995-E07
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- MT-3995 Low group (Experimental)
  Interventions: Drug: MT-3995 Low
- MT-3995 High group (Experimental)
  Interventions: Drug: MT-3995 High
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-3995 Low — MT-3995 Low dose for 8 weeks
  Arms: MT-3995 Low group
Drug: MT-3995 High — MT-3995 High dose for 8 weeks
  Arms: MT-3995 High group
Drug: Placebo — Placebo for 8 weeks
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate pharmacodynamics, safety, tolerability and pharmacokinetics of MT-3995 in Type II Diabetic Nephropathy Subjects with Albuminuria and Moderately Decreased GFR

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type II diabetic nephropathy, who have been treated with angiotensin converting enzyme-inhibitor (ACE-I) or angiotensin II receptor blocker (ARB)
* Glycosylated haemoglobin (HbA1c) ≤10.5%
* An estimated glomerular filtration rate (eGFR) ≥30-<60 mL/min/1.73m^2
* Subject with albuminuria

Exclusion Criteria:

* History of Type I diabetes, pancreas or β-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Serum potassium level <3.5 or >5.0 mmol/L
* Subjects who had acute kidney injury (AKI) within 3 months prior to baseline or have undergone renal dialysis at any time prior to randomisation
* Subjects with a history of renal transplant
* Subjects with clinically significant hypotension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in Urine albumin-to-creatinine ratio (UACR) within group. | up to 8 weeks
Frequency and nature of treatment-emergent adverse events and serious adverse events. | up to 16 weeks

SECONDARY OUTCOMES:
Percentage change from baseline in UACR compared to placebo | up to 8 weeks
Change from baseline in Systolic Blood Pressure and Diastolic Blood Pressure within group. | up to 8 weeks
Plasma concentrations of MT-3995 and its major metabolite | up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (50):
- Bulgaria (7):
  - Investigational site, Blagoevgrad
  - Investigational site, Pazardzhik
  - Investigational site, Pleven
  - Investigational site, Plovdiv
  - Investigational site, Rousse
  - Investigational site, Sofia
  - Investigational site, Varna
- Czechia (8):
  - Investigational site, České Budějovice
  - Investigational site, Český Krumlov
  - Investigational site, Karlovy Vary
  - Investigational site, Ostrava
  - Investigational site, Ostrava-Vitkovice
  - Investigational site, Prague
  - Investigational site, Slaný
  - Investigational site, Znojmo
- Hungary (10):
  - Investigational site, Baja
  - Investigational site, Budapest
  - Investigational site, Debrecen
  - Investigational site, Eger
  - Investigational site, Kistelek
  - Investigational site, Komárom
  - Investigational site, Pécs
  - Investigational site, Szigetvár
  - Investigational site, Szikszó
  - Investigational site, Zalaegerszeg
- Poland (4):
  - Investigational site, Krakow
  - Investigational site, Ruda Śląska
  - Investigational site, Rzeszów
  - Investigational site, Świętochłowice
- Romania (12):
  - Investigational site, Bacau
  - Investigational site, Brăila
  - Investigational site, Bucharest
  - Investigational site, Buzău
  - Investigational site, Cluj-Napoca
  - Investigational site, Deva
  - Investigational site, Iași
  - Investigational site, Oradea
  - Investigational site, Ploiesti, Judet Prahova
  - Investigational site, Satu Mare
  - Investigational site, Târgu Mureş
  - Investigational site, Timișoara
- Slovakia (9):
  - Investigational site, Bardejov
  - Investigational site, Bratislava
  - Investigational site, Levice
  - Investigational site, Lučenec
  - Investigational site, Martin
  - Investigational site, Nitra
  - Investigational site, Prešov
  - Investigational site, Šahy
  - Investigational site, Štúrovo